CLINICAL TRIAL: NCT07244666
Title: Safety and Preliminary Efficacy of a Metabolically Armed Chimeric Antigen Receptor T Cell Therapy Targeting EGFRvIII for Recurrent Glioblastoma
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: META10-EGFRvⅢ-010
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Glioblastoma (GBM)
Keywords: Recurrent glioblastoma; EGFRvIII; metabolically armed; IL-10; CAR-T Cells Therapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Administration of Metabolically Armed EGFRvIII CAR-T cells (Experimental): Patients will be assigned to either the intraventricular injection group or the intravenous injection group, and receive a single infusion of Meta10-EGFRvIII on Day 0.
  Interventions: Drug: Metabolically Armed EGFRvIII CAR-T cells

INTERVENTIONS:
Drug: Metabolically Armed EGFRvIII CAR-T cells — Patients will receive a single infusion of Meta10-EGFRvIII.
  Other Names: Meta10-EGFRvIII; LMC005

SUMMARY:
A Study of Metabolically Armed EGFRvII CAR-T Cells Therapy for Patients With Recurrent Glioblastoma

DETAILED DESCRIPTION:
1. Primary Objective

   Evaluate the safety and efficacy of metabolically armed EGFRvIII CAR-T cell injection in patients with recurrent glioblastoma.
2. Secondary Objectives

Evaluate the pharmacokinetics/pharmacodynamic characteristics of metabolically armed EGFRvIII CAR-T cells in patients with recurrent glioblastoma and the persistence of the CAR-T cells in the subjects.

ELIGIBILITY:
Inclusion Criteria:

* All subjects or their legal guardians must personally sign the written informed consent form approved by the ethics committee in writing before starting any screening procedures;
* Age between 18 and 70 years old (inclusive), both male and female;
* Confirmed diagnosis of recurrent glioblastoma, as specified below:

  1. Previously diagnosed with glioblastoma through histopathological/ molecular pathology reports.
  2. Disease progression or recurrence confirmed by histopathology or imaging (defined as per RANO2.0 criteria as either progression/recurrence or lesions with abnormal enhancement accompanied by hypermetabolism or hyperperfusion changes) that are eligible for use when no standard treatment is available at enrollment;
* Positive EGFRvIII expression detected in tumor cells (confirmed through next-generation sequencing), and only eligible for patients who have previously received EGFRvIII-targeted therapy and relapsed, provided the EGFRvIII remains positive in post-relapse tumor samples;
* Karnofsky Performance Status (KPS) ≥60 points, ECOG score ≤2 (reconfirmed before CAR-T infusion);
* Measurable tumor lesions according to the Response Assessment in Neuro-Oncology (RANO 2.0);
* Adequate peripheral blood obtainable via venipuncture with no contraindications for lymphocyte collection, and sufficient peripheral blood cells collected for CAR-T cell preparation;
* Expected life expectancy ≥12 weeks;
* Adequate organ function (reconfirmed before CAR-T infusion):

  1. Complete blood count [must meet the following criteria within 24 hours prior to whole blood collection: avoid transfusions, platelet transfusions, and colony-stimulating factors (excluding recombinant erythropoietin) within 7 days before testing]:
  2. Blood Biochemistry: Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) ≤2.5 times ULN; serum creatinine ≤1.6 mg/dL; total bilirubin ≤1.5 mg/dL (except for subjects with GBM liver involvement and Gilbert syndrome patients, whose total bilirubin must be <3.0 mg/dL).
  3. Serology: Human immunodeficiency virus (HIV) antibody seronegative. The hepatitis B antigen test is negative, and the hepatitis C antibody test is negative. If the hepatitis C antibody test is positive, reverse transcription polymerase chain reaction (RT-PCR) must be performed to detect the presence of hepatitis B antigen and confirm that the hepatitis C virus (HCV) RNA is negative.
  4. Lung function: normal or grade 1 dyspnea according to CTCAE, SaO2 ≥ 92% in indoor air environment.
  5. Cardiac function: left ventricular ejection fraction (LVEF) ≥40% by echocardiography or radionuclide activity angiography (MUGA) within 1 month of enrollment.
  6. Coagulation function (at least including PT, APTT and INR) is within the normal range.
* Participants using the following medications must meet the following criteria:

  1. Corticosteroids: Treatment doses of corticosteroids must be discontinued 2 weeks prior to starting administration. However, physiological replacement doses of corticosteroids are permitted (hydrocortisone or equivalent <6-12 mg/mm²/day);
  2. At least 8 weeks must have elapsed between completing the last radiotherapy session and initiating treatment;
  3. At least 6 weeks must have passed since the completion of the last nitrosourea-based chemotherapy regimen;
  4. At least 14 days must have elapsed since the completion of the last temozolomide or other chemotherapy regimens before treatment initiation. If the subject has recently received targeted therapy and adverse events related to their targeted drug have resolved to baseline levels, screening may begin after a 2-week washout period (for bevacizumab, a total of 4 weeks of washout is required after confirming no bleeding caused by gastrointestinal ulcers). For long-term chronic low-grade (≤2) adverse events such as paronychia, eligibility will be determined by the investigator.
* The investigator determines that the subject has recovered from toxicity caused by prior anti-tumor treatment to grade 1 or below (except for special grade 2 or below toxicity that could not be recovered in a short period of time, such as hair loss), and is suitable for pre-treatment chemotherapy and CAR-T cell therapy.
* All male subjects and women of childbearing age must agree to use highly effective contraceptive methods for at least 12 months after LMC005 infusion until two consecutive PCR tests show no residual CAR-T cells in the body.
* Patients in the intraventricular injection group must additionally meet the following criteria: The investigator determines that the intracranial tumor is suitable for Ommaya sac implantation.

Exclusion Criteria:

* Subjects exhibiting other severe central nervous system disorders deemed by the investigator to be unrelated to the indication;
* Subjects anticipated to require systemic corticosteroid use within three months due to disease progression related to the indication;
* Subjects who have received the following medications:

  1. Corticosteroids at therapeutic doses (defined as prednisone >20 mg/day, hydrocortisone >20 mg/day, methylprednisolone >4 mg/day, dexamethasone >0.75 mg/day, betamethasone >0.5 mg/day) within 7 days prior to leukapheresis or within 72 hours before CAR-T cell administration;
  2. Lymphocyte-toxic chemotherapy (e.g., cyclophosphamide, ifosfamide, bendamustine) administered within 2 weeks prior to leukapheresis;
  3. Investigational drugs from other clinical trials used within 4 weeks prior to blood collection. Exception: Patients whose prior trial medications were ineffective or whose disease progressed during the trial, provided at least 3 half-lives have elapsed since the last dose before leukapheresis;
  4. Radiotherapy received within 4 weeks prior to blood collection.
* Subjects with active hepatitis B (defined as hepatitis B surface antigen positivity or core antibody positivity with HBV DNA >1000 copies/mL) or active hepatitis C (HCV RNA positive);
* Subjects testing positive for HIV antibodies or Treponema pallidum antibodies;
* Subjects with uncontrolled acute life-threatening bacterial, viral, or fungal infections (e.g., positive blood culture ≤72 hours prior to LMC005 infusion);
* Subjects with unstable angina and/or myocardial infarction within 6 months prior to signing informed consent; or subjects with severe stroke or deep venous thrombosis (DVT) within 12 months prior to signing informed consent;
* Subjects with a history of or concurrent malignant tumors, except those meeting the following criteria:

  1. Surgically excised non-melanoma skin cancer;
  2. Curatively treated carcinoma in situ of the cervix;
  3. Localized prostate cancer;
  4. Low-stage bladder cancer;
  5. Ductal carcinoma in situ of the breast;
  6. Malignancies without recurrence or treatment within the past 2 years.
* Pregnant or lactating female subjects (women of childbearing potential with a positive pregnancy test result during screening);
* Subjects with active autoimmune diseases (e.g., Guillain-Barré syndrome, systemic lupus erythematosus);
* Subjects with a history of QT interval prolongation or other significant cardiac diseases;
* Subjects with contraindications to MRI scanning, including embedded metallic materials/devices (e.g., pacemakers);
* Other circumstances identified by the investigator as rendering the subject unsuitable for this study (e.g., poor compliance).

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | up to 12 months
  To characterize the safety profile of Meta10-EGFRvIII in patients with recurrent glioblastoma as assessed by incidence of adverse events. Adverse events will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 months after receiving the first dose of CAR-T cell infusion
  To evaluate the proportion of participants who have a confirmed partial response (PR) and complete response (CR) per RANO2.0 as assessed by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Chongran Sun, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No